CLINICAL TRIAL: NCT05241262
Title: A Multiple Ascending Phase 1 Dose Study of N-acetylcysteine in the Treatment of Patients With the m.3243A>G Mutation and Low Brain Glutathione Levels
Brief Title: Study of N-acetylcysteine in the Treatment of Patients With the m.3243A>G Mutation and Low Brain Glutathione Levels
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Michio Hirano, MD (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Michio Hirano, MD, Lucy G. Moses Professor of Neurology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAT7415; PR 190511 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-02-03; First posted 2022-02-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Mitochondrial Disease
Keywords: m.3243A>G; MELAS; diabetes; deafness
MeSH Terms: conditions — Mitochondrial Diseases; MELAS Syndrome; Diabetes Mellitus; Deafness | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: 18 Carrier relatives will participate in a dose finding study of NAC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active drug (NAC) (Experimental): Participants will receive NAC for 3 months.
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — 1800, 3600 or 5400 mg NAC per day (divided into 3 daily doses) depending on dose toxicity plan
  Other Names: NAC

SUMMARY:
N-Acetylcysteine (NAC), an anti-oxidant, will be studied to investigate the effects on brain glutathione levels, cognitive skills, motor skills, and quality of life.

A group of 18 participants will take either 1800, 3600 or 5400 mg per day of N-acetylcysteine (NAC) for 3 months in this dose escalation study. The investigators want to determine first if the 3600 mg dose per day is safe and might provide some efficacy. If the 3600 mg dose is safe, then additional participants will be treated with 5400 mg per day of NAC, for up to a total of 18 participants. If the 3600 mg per day dose is unsafe, then participants will be treated with the 1800 mg per day dose. Data from this pilot study will be used to determine the most safe and effective dose of NAC for a future clinical trial.

DETAILED DESCRIPTION:
Patients with the m.3243A>G mitochondrial mutation often have low brain glutathione levels. These low levels can reduce the repair processes in the brain to fix toxic chemicals that result from a mitochondrial disorder. The investigators are aware of a potent anti-oxidant, called N-Acetylcysteine (NAC), that may improve the brain glutathione level when taken in sufficient quantity. In turn, cognitive and motor skill impairment may improve as these toxic levels are reduced. will be studied to investigate the effects on brain glutathione levels, cognitive skills, motor skills, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80 years
* Low brain glutathione (GSH) levels as determined by magnetic resonance spectroscopic imaging (MRSI)
* Individuals who carry, or are suspected of carrying the m.3243A>G mitochondrial mutation (genetic confirmation of mutation required prior to initiation of NAC)

Exclusion Criteria:

* Individuals with normal brain glutathione levels
* Pregnant or lactating individuals
* Medically unstable as determined by the Principal Investigator
* Allergy to NAC or other sulfur-containing drug
* Inability to adhere to study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of NAC | 4 months
  Establish maximum tolerated dose of NAC by initiating dosing at one level, then increasing or decreasing dose based on toxicity. The MTD is defined as the dose associated with a target probability of dose limiting toxicity (DLT) of 0.10.

SECONDARY OUTCOMES:
Columbia Neurological Score | 4 months
  The Columbia Neurological Score evaluates patients with cerebral energy failure syndromes and quantifies key neurological examination domains. The Columbia Neurological Score ranges from 0 to 76 with higher scores indicating less clinical severity.
Change in Global Neuropsychological Score | 4 months
  A composite global neuropsychological score is used to assess loss of cognitive function. The global neurological score is derived from measures across a standard neuropsychological battery. Test domains include: Memory, Orientation, Abstract reasoning, Dementia,Language,Word Association, and Naming. The scores range from 0 to 2 with higher scores indicating worsening cognitive function.
Change in Functional Exercise Capacity (6 minute walk test (6MWT)) | 4 months
  The 6MWT is an objective evaluation of functional exercise capacity assessing the distance a person can walk in six minutes.
Change in Karnofsky Performance Scale (KPS) Score | 4 months
  KPS assesses functional activities of daily living (ADL). Scores range from 0 to 100 with a score of 0 defined as death and 100 defined as normal; no complaint; no evidence of disease (better outcome).
Change in Brain glutathione (GSH) level | 4 months
  As measured by brain Magnetic resonance Imaging and Magnetic resonance spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No